CLINICAL TRIAL: NCT04114747
Title: Impact of Continuous Renal Replacement Therapy on Renal Oxygenation, Blood Flow and Function
Brief Title: Renal Physiology During Continuous Renal Replacement Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Kristina Svennerholm, Principal investigator, MD, PhD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Kidney and dialysis
Record Dates: First submitted 2019-09-23; First posted 2019-10-03 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: AKI; Continuous Renal Replacement Therapy; Dialysis; Intensive Care; Renal Blood Flow; Renal Failure; Blood Pressure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: To describe renal physiology parameters when starting CRRT and compare renal physiology parameters when using high blood pressure target (MAP 80-90 mmHg) and low blood pressure target (MAP 60-70 mmHg).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Starting at high blood pressure (Experimental): Patients in this arm are randomized to have high target blood pressure at MAP 80-90 mmHg during the first recordings, thereafter they will receive low blood pressure target 60-70 mm Hg
  Interventions: Other: Starting at high or low blood pressure
- Starting at low blood pressure (Experimental): Patients in this arm are randomized to have low target blood pressure at MAP 60-70 mmHg during the first recordings, thereafter they will receive high blood pressure target 80-90 mm Hg
  Interventions: Other: Starting at high or low blood pressure

INTERVENTIONS:
Other: Starting at high or low blood pressure — Using norepinephrine, patients will receive high or low blood pressure to start with and after measurements cross to receive the other blood pressure target

SUMMARY:
Approximately 50% of patients in the intensive care unit (ICU) develop acute kidney injury (AKI) and more than 10% need dialysis. There is no treatment for AKI. Care is aiming for optimization of circulation and blood flow to the kidneys and avoiding nephrotoxic agents.

There is conflicting data concerning whether early or late dialysis is harmful for the kidneys. No one has examined the physiological changes in the kidney when starting dialysis and which blood pressure that leads to most optimal physiological conditions for the kidneys during dialysis. In this descriptive study of 20 ICU patients suffering from AKI we aim to investigate renal physiology when starting continuous renal replacement therapy (CRRT) and also at different target blood pressures using retrograde renal vein thermodilution technique. In parallel we will also investigate and validate this invasive method with contrast enhanced ultrasound of the kidneys.

ELIGIBILITY:
Inclusion Criteria:

AKI, according to KDIGO, stage 2 or 3 but with preserved urine production. Treated in the ICU at Sahlgrenska University Hospital Written, signed informed consent Male and female subjects ≥18 years

Exclusion Criteria:

Emergency need for dialysis Allergy to contrast media (used for CEUS)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Renal blood flow and CRRT | 6 hours
  Changes in renal blood flow when CRRT is started? How will renal blood flow and oxygenation change at different blood pressure targets?
Renal blood flow and blood pressure | 6 hours
  Renal blood flow changes at different mean arterial blood pressure targets during CRRT?
Glomerular filtration rate (GFR) and blood pressure | 6 hours
  GFR changes at different mean arterial blood pressure targets during CRRT?
Glomerular filtration rate (GFR) and CRRT | 6 hours
  Changes in GFR when CRRT is started?
Renal oxygenation during CRRT | 6 hours
  Renal oxygenation before CRRT and during CRRT
Renal oxygenation and blood pressure | 6 hours
  Renal oxygenation changes at different mean arterial blood pressure targets during CRRT?

SECONDARY OUTCOMES:
Contrast enhanced renal ultrasound (CEUS) | 2 hours
  Validation of CEUS compared to retrograde renal vein thermodilution in measuring renal blood flow
atrial natriuretic peptide (ANP) | 6 hours
  Differences in serum atrial natriuretic peptide (ANP) during CRRT

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Svennerholm, MD PhD, Principal Investigator
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No